CLINICAL TRIAL: NCT01195558
Title: Development of a Patient Registry of Blind Subjects With Sleep-related Problems
Brief Title: Patient Registry of Blind Subjects With Sleep-related Problems
Status: Recruiting | Type: Observational
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00005099
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Sleep-wake Disorder in Blind Individuals
Keywords: Non-24; N24HSWD; Blindness; Sleep; Wake; Circadian Rhythm; Nap
MeSH Terms: conditions — Blindness | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blind with sleep problems: Blind individuals with no light perception and with sleep-related problems who may suffer from Non-24
  Interventions: Other: Data collection on blindness and sleep problems

INTERVENTIONS:
Other: Data collection on blindness and sleep problems — Data related to degree of vision impairment and sleep problems is collected through a phone or web survey
  Other Names: Data Collection

SUMMARY:
Non-24-hour sleep-wake disorder (Non-24) is a condition experienced primarily by totally blind individuals that results in abnormal night sleep patterns and chronic daytime sleepiness. This is a research protocol to develop a patient registry of subjects who may suffer from Non-24 and who are blind. Subjects participate in the study through a phone survey. This registry will be used to better understand, sleep related problems in blind individuals, including the investigation of a potential treatment, recruitment for future clinical studies, and to provide a forum for raising awareness about Non-24. The survey consists of questions regarding the degree of vision impairment and sleep problems that the subjects may be experiencing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or legal guardians must be at least 18 years of age to participate in the telephone survey. Parents or legal guardians may represent children from 0 through 17 years who meet the following criteria.
2. Subjects must be blind.
3. Subjects must have some self-described problem with sleep or daytime sleepiness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population of blind individuals
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-04; Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Number of blind participants | ongoing

SECONDARY OUTCOMES:
Sleep/wake disruptions | ongoing

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Pharmaceuticals, Washington D.C., District of Columbia, United States